CLINICAL TRIAL: NCT01699464
Title: Phase 2b Dose-response of AR-12286 in Patients With Elevated Intraocular Pressure for 3 Months
Brief Title: A Study Assessing the Safety and Ocular Hypotensive Efficacy of AR-12286 in Patients With Elevated Intraocular Pressure for 3 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR-12286-CS206
Record Dates: First submitted 2012-10-02; First posted 2012-10-03 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Ocular Hypertension; Open-angle Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AR-12286 Ophthalmic Solution 0.7% (Experimental): AR-12286 Ophthalmic Solution 0.7%, both eyes
  Interventions: Drug: AR-12286 Ophthalmic Solution 0.7%
- AR-12286 Ophthalmic Solution 0.5% (Experimental): AR-12286 Ophthalmic Solution 0.5% both eyes
  Interventions: Drug: AR-12286 Ophthalmic Solution 0.5%
- Timolol maleate ophthalmic solution 0.5% (Active Comparator): Timolol maleate ophthalmic solution 0.5% both eyes
  Interventions: Drug: Timolol maleate ophthalmic solution 0.5%

INTERVENTIONS:
Drug: AR-12286 Ophthalmic Solution 0.7% — Ophthalmic Solution
  Arms: AR-12286 Ophthalmic Solution 0.7%
Drug: AR-12286 Ophthalmic Solution 0.5% — Ophthalmic Solution
  Arms: AR-12286 Ophthalmic Solution 0.5%
Drug: Timolol maleate ophthalmic solution 0.5% — Ophthalmic Solution
  Arms: Timolol maleate ophthalmic solution 0.5%

SUMMARY:
A double-masked, parallel study of AR-12286 Ophthalmic Solution 0.5%, or 0.7% (q.d., PM) or timolol maleate Ophthalmic Solution, 0.5% (b.i.d.), O.U. for 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. 18 year of age or greater. (India_ Maximum age of 65 years)
2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT).
3. Unmedicated (post-washout) IOP ≥ 24 mm Hg at 2 eligibility visits (0800 hr), 2-7 days apart, and ≥ 22 mm Hg at 1000 and 1600 hrs at the second qualification visit. If only one eye meets the IOP criteria it must be the same eye that met the criteria at all the qualification timepoints.
4. Corrected visual acuity in each eye +1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200).
5. Able and willing to give signed informed consent and follow study instructions.

Exclusion Criteria:

Ophthalmic

1. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure or narrow angles. Note: Previous laser peripheral iridotomy is NOT acceptable.
2. IOP > 36 mm Hg
3. Current use of more than 1 ocular hypotensive medications (Note: fixed dose combinations are considered multiple medications).
4. Known hypersensitivity to any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics.
5. Previous glaucoma intraocular surgery or glaucoma laser procedures in study eye(s).
6. Refractive surgery in study eye(s) (e.g., radial keratotomy, PRK, LASIK, etc.).
7. Ocular trauma within the past six months, or ocular surgery or laser treatment within the past three months.
8. Evidence of ocular infection, inflammation, clinically significant blepharitis or conjunctivitis at baseline (Visit 1), or a history of herpes simplex keratitis
9. Ocular medication of any kind within 30 days of Visit 1, with the exception of a) ocular hypotensive medications (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after Visit 1) or c) lubricating drops for dry eye (which may be used throughout the study).
10. Clinically significant ocular disease (e.g. uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe (i.e., cup-disc ratio > 0.8).
11. Central corneal thickness greater than 600 µm.
12. Any abnormality preventing reliable applanation tonometry of either eye.

    Systemic:

    Systemic:
13. Clinically significant abnormalities (as determined by the treating physician) in laboratory tests at screening.
14. Known hypersensitivity or contraindication to beta adrenoceptor antagonists including chronic obstructive pulmonary disease or bronchial asthma; abnormally low blood pressure or heart rate; second or third degree heart block or congestive heart failure; severe diabetes).
15. Clinically significant systemic disease (e.g., myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
16. Participation in any investigational study within the past 30 days.
17. Changes of systemic medication that could have a substantial effect on IOP within 30 days prior to screening, or anticipated during the study.
18. Due to the current status of the preclinical safety program, women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Mean IOP across subjects within treatment group at each post-treatment timepoint of Month 3 | Month 3
  Intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Brian Levy, OD, Study Director — Aerie Pharmaceuticals, Inc.